CLINICAL TRIAL: NCT02341924
Title: Validating the "Foods for Health" Portfolio of Functional Food Products: Effects on Lipid and Blood Glucose Management in Individuals Intolerant of Statin (HMG-CoA Reductase Inhibitor) Therapy
Brief Title: Validating the "Foods for Health" Portfolio of Functional Food Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Agri-Health Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: B2014:113
Record Dates: First submitted 2014-12-10; First posted 2015-01-19 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2021-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Portfolio of functional foods (Experimental): A portfolio of functional foods provided as packaged shelf-stable food products (Step One Treatment) which will include foods such as oatmeal, pancakes, cranberry bars, chocolate bars, smoothies, and a sprinkle offering which can be added to almost any food to enhance its nutritional impact.
  All products are interchangeable in terms of their nutrients of interest and contain a minimum of 5 g of fibre, 1800 mg of omega-3 fatty acids, 1000 mg of phytosterols and 1800 µmol antioxidants per serving. Calorie counts range from 110-190 kcal per serving.
  Interventions: Other: Portfolio of functional foods
- Control foods (Placebo Comparator): Control products will be like-items drawn from the general grocery marketplace. Test and control products will be packaged and coded identically.
  Interventions: Other: Control foods

INTERVENTIONS:
Other: Portfolio of functional foods
  Arms: Portfolio of functional foods
Other: Control foods
  Arms: Control foods

SUMMARY:
The objective of this research project is to investigate the ability to affect cardiovascular disease (CVD) risk factors through a novel, easily implemented functional food-based approach. The goal of the proposed project is to evaluate the effect of a range of proprietary products specifically formulated to deliver convenient pre-packaged condition-specific foods to positively impact blood cholesterol levels in statin intolerant and/or statin unwilling participants. The specific aim of this project is to evaluate the changes in serum low-density lipoprotein (LDL)-cholesterol, triglyceride (TG) glucose, insulin and high-sensitivity C-reactive protein (hsCRP) concentrations over a 4 week regimen using healthy tasty foods which are self-selected by a statin intolerant patient group.

ELIGIBILITY:
Inclusion Criteria:

Participants aged > 21 to < 65 years will be recruited on the basis of ability to give informed consent and being unwilling to use or intolerant of at-least one statin medication.

Exclusion Criteria:

Participants will be excluded if they are unable to speak/read in English or are unable or unwilling to temporarily hold all statin/lipid lowering therapies including supplements throughout the study period.

Participants with diabetes or severe obesity (body mass index, BMI, > 35 kg/m2) will be excluded.

Women who are pregnant or planning to be pregnant during the study period will not be eligible for the study.

Participants with any food allergies/intolerances, food restrictions due to medical, religious or philosophical reason - including Kosher, vegan, vegetarian, high protein, low-carbohydrate, low-phosphorus, etc. other than attempting to follow an eating plan as generally advocated by the American Heart Association (low sodium, low cholesterol, reduced fat, etc.) will be excluded.

Participants will not be eligible if their baseline fasting LDL-C is < 100 mg/dL or > 190 mg/dL; or evidence of tissue cholesterol deposition; if their baseline fasting TG is > 400 mg/dL or baseline fasting blood glucose is > 126 mg/dL.

Consumption of more than 2 alcoholic drink/day or history of alcoholism or drug dependence will also serve as an exclusion criterion.

Smokers will be excluded from the study.

History of non-skin cancer, history of melanoma, history of rheumatoid arthritis or other chronic rheumatologic condition, history of advanced cardiovascular disease (moderate or greater valvular disease, history congestive heart failure, known coronary artery disease, history dysrhythmias requiring medical or surgical intervention), , known chronic liver or renal disease, diabetes, inflammatory bowel disease, celiac disease, uncontrolled thyroid disease, hormonal supplementation(other than thyroid), pancreatitis, gallbladder or biliary disease, neurological/psychological disease, and gastrointestinal disorders that could interfere with fat absorption will be excluded.

Individuals with uncontrolled hypertension having systolic blood pressure >150 mm Hg or diastolic blood pressure >100 mm Hg will be excluded from the study.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Change in fasting serum lipids (total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol and triglycerides) | Baseline (days 1 and 2) and Endpoint (days 29 and 30)

SECONDARY OUTCOMES:
Change in fasting serum glucose | Baseline (days 1 and 2) and Endpoint (days 29 and 30)
  Homeostasis model of assessment for insulin resistance (HOMA-IR) index will also be calculated
Change in fasting insulin | Baseline (days 1 and 2) and Endpoint (days 29 and 30)
  Homeostasis model of assessment for insulin resistance (HOMA-IR) index will also be calculated
Change in fasting C-reactive protein | Baseline (days 1 and 2) and Endpoint (days 29 and 30)

CONTACTS AND LOCATIONS:
Overall Officials: Rotimi E Aluko, PhD, Principal Investigator — University of Manitoba, Richardson Centre for Functional Foods and Nutraceuticals
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Kopecky SL, Alias S, Klodas E, Jones PJH. Reduction in Serum LDL Cholesterol Using a Nutrient Compendium in Hyperlipidemic Adults Unable or Unwilling to Use Statin Therapy: A Double-Blind Randomized Crossover Clinical Trial. J Nutr. 2022 Feb 8;152(2):458-465. doi: 10.1093/jn/nxab375. PMID 35079806